CLINICAL TRIAL: NCT04008810
Title: Serum Neutrophil Gelatinase-associated Lipocalins (NGAL) Ability to Predict Chronic Kidney Disease and the Number of Readmissions in Patients Admitted in the Emergency Department - a Longitudinal Prospective Study
Brief Title: Serum Neutrophil Gelatinase-associated Lipocalins (NGAL) and Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Hillerod Hospital, Denmark (Other)
Collaborators: BioPorto Diagnostics (Industry)
Responsible Party: Principal Investigator, Vicky Jenny Rebecka Wetterstrand, Principal Investigator and Physician, Nordsjaellands Hospital
Other Study IDs: H-19003424
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Diseases; CKD; NGAL; Neutrophil Gelatinase-associated Lipocalin; Emergency Department; AKI; Acute Kidney Injury
Keywords: renal insufficiency; renal failure; acute kidney injury; AKI
MeSH Terms: conditions — Renal Insufficiency, Chronic; Emergencies; Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute kidney injury (AKI) is associated with significant morbidity and mortality, and because no specific treatment is available, early acknowledgment is needed. The incidence of AKI and chronic kidney disease (CKD) have been increasing over time but it is not until the past decade there is an understanding of a bidirectional nature between AKI and CKD, where AKI predisposes to CKD and vice versa. The criteria for diagnosing AKI is through serum creatinine (sCr) and/or urine output. As detection of sCr-increases are delayed by 48-72 hours it is not an optimal biomarker for early recognition of AKI. In contrast the biomarker neutrophil gelatinase-associated lipocalin (NGAL) has shown to predict AKI within 12h of critical disease or postoperative, and without the requirement of prior measurements for comparison.

The purpose of the project is to investigate if the relatively new biomarker NGAL (neutrophil gelatinase-associated lipocalin), which is known to be able to detect AKI in an early phase, can be used to detect development of CKD and potential future hospital admissions in a relatively large and diverse cohort of patients admitted to the Acute Emergency Department at North Zealand Hospital.

The study is designed as a longitudinal prospective study where there is an enrollment estimation of 3600 unselected patients over one year. Blood tests will be taken when admitted and thereafter every day for the first week and subsequently every once a week throughout hospitalization. Patients that are sent home the same day, will still be included in the study but without further NGAL analyses.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is associated with significant morbidity and mortality, and because no specific treatment is available, early acknowledgment is needed. The incidence of AKI and chronic kidney disease (CKD) have been increasing over time but it is not until the past decade there is an understanding of a bidirectional nature between AKI and CKD, where AKI predisposes to CKD and vice versa. The criteria for diagnosing AKI is through serum creatinine (sCr) and/or urine output. As detection of sCr-increases are delayed by 48-72 hours it is not an optimal biomarker for early recognition of AKI. In contrast the biomarker neutrophil gelatinase-associated lipocalin (NGAL) has shown to predict AKI within 12h of critical disease or postoperative, and without the requirement of prior measurements for comparison.

The purpose of the project is to investigate if the relatively new biomarker NGAL (neutrophil gelatinase-associated lipocalin), which is known to be able to detect AKI in an early phase, can be used to detect development of CKD and potential future hospital admissions in a relatively large and diverse cohort of patients admitted to the Acute Emergency Department at North Zealand Hospital.

The study is designed as a longitudinal prospective study where there is an enrollment estimation of 3600 unselected patients over one year. Blood tests will be taken when admitted and thereafter every day for the first week and subsequently every once a week throughout hospitalization. Patients that are sent home the same day, will still be included in the study but without further NGAL analyses. There will be follow-up time in all patients included in the study, up to one year after admission through the Danish National Patient Register and medical journals to see if the patients are reinstated, what they are diagnosed with and if they have had other hospital contacts. This will further be done to examine if NGAL is better at predicting the number of hospital contacts, up to one year after discharge.

Primary endpoint:

If NGAL can predict development of CKD defined as eGFR < 60ml/min per 1.73 m^2 and/or albumin/creatinine ratio >= 30mg/g over 3 months in patients upfilling the AKI criteria with a delta-creatinine >= 26,5 umol/l during the initial hospital admission, within one year from first admission. Cystatin C values will be compared to NGAL.

Secondary endpoints:

* The risk assessments (risk factor and risk patients) described by The Danish Society of Nephrology will be operationalized and interpreted. The data will be collected from medical records, Danish National Patient Registry (DNPR) and Danish Register of Causes of Death (DRCD) in patients with AKI.
* Patients meeting >= 1 of the either "risk factors" or "risk patients" in risk of developing AKI and with a delta-creatinine >=26,5 l mol/L and/or an sCr increase by 50% in seven days during the primary hospital stay, will be compared with NGAL and information from medical records, hospital discharge diagnosis, DNPR and DRCD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and
* Male or female aged >= 18 years and
* Admitted to the ED at North Zealand University Hospitals, on one of the three chosen days of the month
* At least one valid delta-creatinine

Exclusion Criteria:

* Admitted through pediatric-, gynecologic-, obstetric department and intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unselected patients admitted through the emergency department
Sampling Method: Probability Sample
Enrollment: 1032 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Development of chronic kidney disease (CKD) | up to one year from first admission
  Neutrophil Gelatinase-associated Lipocalin (NGAL) in ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- North Zealand Hospital, Hillerød, Denmark